CLINICAL TRIAL: NCT03966313
Title: Perioperative Modification of Hemostasis During Ventricular Assist Device Implantation
Acronym: HemostVAD
Status: Terminated | Type: Observational
Why Stopped: Due to inclusion difficulties following the evolution of surgical indications, which were clearly restricted, making patient inclusion too complex.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7287
Record Dates: First submitted 2019-05-17; First posted 2019-05-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: End-stage Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Whole blood
  * Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: ventricular assist device implantation — Blood sampling in patients under surgery for ventricular assist device implantation at five time points:
  * After anesthetic induction
  * Before starting the device
  * 2h, 6h and 48h after starting the device

SUMMARY:
Implanting a ventricular assist device (VAD) is a promising therapy for end-stage cardiac failure. However, the implantation of these devices is associated with a high risk of severe hemorrhages and massive blood product transfusion in the first 48 hours following the implantation. The primary purpose of this study is to assess the functionality of the von Willebrand Factor (vWF) which is essential for hemostasis. The hypothesis is that the high shear stress generated by these VAD expose ADAMTS13 cleaving site on the vWF. This result in a loss of high molecular weight vWF and an acquired von Willebrand syndrome.

The secondary purpose of the protocol is to assess platelet function after the implantation of VAD. Indeed, platelet function might be affected shortly after the implantation of the device.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Who gave his consent to the study
* With an end-stage heart-failure
* Under surgery for a ventricular assist device implantation
* Scheduled or in emergency

Exclusion Criteria:

* Preoperative anemia less than 7 g/dL
* Subject under the protection of justice
* Subject under guardianship or curatorship
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with end-stage heart failure (acute or chronic) under surgery for implantation of a ventricular assist device.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

PRIMARY OUTCOMES:
Von Willebrand Factor activity | From Baseline to 48 hours
  Change of Von Willebrand Factor from Baseline to 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaire de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No